CLINICAL TRIAL: NCT00114582
Title: Optimizing the Ambiance During Mealtimes in Dutch Nursing Homes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2420.0021
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Malnutrition
Keywords: family style dinner; quality of life; nutritional status; nursing home residents
MeSH Terms: conditions — Malnutrition

INTERVENTIONS:
Procedure: family style dinner

SUMMARY:
Optimizing the social and physical ambiance during mealtimes in Dutch nursing homes: implementation and evaluation of the effect with respect to quality of life, nutritional status and physical performance.

DETAILED DESCRIPTION:
Study design: During six months the intervention group had their meals in family style, and the control group received the usual tray services.

Hypothesis: We hypothesized that the intervention program had a positive effect on quality of life, food intake, body weight, physical performance, and biochemical data (hematocrit, hemoglobin, leucocytes, ferretin, albumin, homocysteine and folate) among the residents in the intervention group, while these outcome measures would regularly decline among the residents in the control group.

Site and participants: Nursing homes volunteered to participate in the study. In each nursing home there was a control and intervention ward. Only residents with a chronic somatic disorder were included. Residents were excluded when they were in a terminal phase of a disease, had total parenteral feeding or were not able to give informed consent due to their physical or mental condition. The ethical committee and the client board of the nursing homes and the medical ethical committee of Wageningen University approved the study protocol.

Intervention: The intervention program lasted for six months and was based on an inventory research of mealtime ambiance models in the Netherlands. The program consisted of five aspects: table dressing, food services, staff protocol, residents' protocol, and mealtime protocol. Before the start of the meal, tables were set with tablecloths, full cutlery and plates. The cooked meal was served in dishes and residents had the opportunity to choose between two kinds of vegetables, two kinds of meat and potatoes.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home residents with a chronic somatic disease and long term care

Exclusion Criteria:

* Residents were excluded when they were in a terminal phase of a disease, had total parenteral feeding or were not able to give informed consent due to their physical or mental condition.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-04; Study Completion 2003-12

PRIMARY OUTCOMES:
Nutritional status
Quality of life
Physical performance

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Background] Mathey MF, Vanneste VG, de Graaf C, de Groot LC, van Staveren WA. Health effect of improved meal ambiance in a Dutch nursing home: a 1-year intervention study. Prev Med. 2001 May;32(5):416-23. doi: 10.1006/pmed.2001.0816. PMID 11330991
- [Background] Nijs K, Vanneste V, de Graaf K, van Staveren W. [Project models to improve the ambiance during meal times in Dutch nursing homes: incentives and barriers for implementation]. Tijdschr Gerontol Geriatr. 2003 Dec;34(6):246-53. Dutch. PMID 15007956
- [Result] Nijs KA, de Graaf C, Kok FJ, van Staveren WA. Effect of family style mealtimes on quality of life, physical performance, and body weight of nursing home residents: cluster randomised controlled trial. BMJ. 2006 May 20;332(7551):1180-4. doi: 10.1136/bmj.38825.401181.7C. Epub 2006 May 5. PMID 16679331